CLINICAL TRIAL: NCT00037804
Title: Irinotecan in Treating Patients With Refractory Solid Tumors and Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Purpose: Treatment
Other Study IDs: M64750017; NCT00002958 (obsolete NCT alias)
Record Dates: First submitted 2002-05-21; First posted 2002-05-22 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Unspecified Adult Solid Tumor; Chemotherapy; Liver Dysfunction; Neoplasms, Solid Tumor
Keywords: Pharmacia
MeSH Terms: conditions — Liver Diseases; Neoplasms | interventions — Irinotecan

INTERVENTIONS:
Drug: Irinotecan

SUMMARY:
Drugs used in chemotherapy us different ways to stop tumor cells from dividing so they stop growing or die. Irinotecan may be effective in treating patients with refractory solid tumors and liver dysfunction.

ELIGIBILITY:
Other specific inclusion/exclusion criteria may apply. In order to determine eligibility, further examination by the investigator is necessary.

Inclusion Criteria: Histological proof of malignant solid tumor that is refractory to standard forms of therapy or for which no known curative therapy exists; Measurable or evaluable disease; At least 6 weeks since prior chemotherapy with nitrosoureas; At least 28 days since prior anticancer therapy and recovered; At least 4 weeks since prior radiation therapy and recovered; Age 18 years or older; SWOG 0-2; Life expectancy of at least 12 weeks; Segmented neutrophils with bands at least 1,500/mm3; Hemoglobin at least 9.0 g/dL and platelet count at least 100,000/mm3; Prothrombin time and partial thromboplastin time no greater than 2.0 times control; INR no greater than 3.0 times control; Concurrent use of coumadin allowed only if dose is stable and prothrombin time and INR is stable; Total serum bilirubin at least 1.5 but no greater than 5.0 times upper limit of normal; SGOT/SGPT no greater than 5 times upper limit of normal; SGOT/SGPT at least 1.5 but no greater than 20.0 times upper limit of normal; Creatinine no greater than 2

Exclusion Criteria: Patients expressing tumor markers as their only evidence of disease or who have previously irradiated areas that have not increased in size; Prior chemotherapy treatment with irinotecan and mitomycin; Prior abdominal and/or pelvic radiation therapy; Current history of hepatitis B infection or positive test for hepatitis B surface antigen; Hepatic encephalopathy including somnolence, confusion, or asterixis; History of myocardial infarction within 6 months or history of congestive heart failure (CHF); clinical evidence of CHF; Evidence of arrhythmia in patients with history of cardiac arrhythmia; Uncontrolled hypertension, unstable angina, active CHF, or serious uncontrolled cardiac arrhythmia; Interstitial pneumonia or fibroid lung (patients must have large pleural effusions drained and sclerosed or controlled prior to study; patients must have clinically apparent ascites drained prior to irinotecan treatment); CNS metastases or carcinomatous meningitis; Concurrent use of anticonvulsants; Active or uncontrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Center, Detroit, Michigan
  - Research Center, New Brunswick, New Jersey
  - Research Center, Nashville, Tennessee
  - Research Center, Marshfield, Wisconsin